CLINICAL TRIAL: NCT05960916
Title: Primary Stability of Immediate Dental Implant Using Osseodensification and Conventional Burs (A Randomized a Clinical Comparative Prospective Study)
Brief Title: Primary Stability of Immediate Implant Using Versah Versus Conventional Burs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mustafa Thamer Naji, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 121189
Record Dates: First submitted 2023-07-02; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Edentulous Alveolar Ridge
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Dividing two groups according drill type and parallelly measured during study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Densah® bur (Experimental): Densah is a bur that used for drilling of the alveolar ridge that have low bone density, narrow alveolar ridge, and sinus lifting procedure in dental implant preparation technique.
  Interventions: Procedure: Densah® burs
- Conventional bur (Active Comparator): Conventional bur is the gold standard bur that used to prepare the osteotomy for dental implant.
  Interventions: Procedure: Conventional Burs

INTERVENTIONS:
Procedure: Densah® burs — Osseodensification is a non-excavating implant site preparation technique, it creates a densified layer of surrounding bone through compaction autografting while simultaneously plastically expanding the bony ridge at the same time facilitating for placement of large diameter implants and also avoiding fenestration and dehiscence defects.
  Other Names: Study group
  Arms: Densah® bur
Procedure: Conventional Burs — Conventional burs is the gold standard that used to prepare the osteotomy site by drilling of the bone and creating a bed for implant placement, it is used according to the manufacturer instructions.
  Other Names: Control group
  Arms: Conventional bur

SUMMARY:
This study is designed as a Prospective Randomized Clinical Trail, Evaluate the effect of osseodensification technique on primary stability in comparison to the conventional drilling technique in immediate single fresh extraction sockets.

DETAILED DESCRIPTION:
In this study, 30 dental implants inserted immediately after tooth extraction (not a multi-rooted tooth) as a two groups according to bur drill technique and measure the primary stability by osstell devise based on resonance frequency analysis (RFA) value which is scaled from 1-100, after 16 weeks measuring the secondary stability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and medically fit patients
* Patients age ≥18 years for both gender
* Apical bone ≥ 2mm from vertical structure showed in x-rays.
* Patient has tooth or teeth with single root anterior and\or posterior area cannot
* restored by another dental treatment procedure.

Exclusion Criteria:

* Patient with active periodontal disease.
* Pregnancy or lactation.
* A local or systemic disorder that is contraindicated for the minor surgical procedure
* and may affect healing process.
* Any irradiation in head and neck area.
* Heavy smoking habit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary Implant Stability Quotient (ISQ) | baseline value of implant stability measured immediately after implant installation (primary stability)
  immediately after implant placement the ISQ value measured by RFA device (Osstell)

SECONDARY OUTCOMES:
Secondary Implant Stability Quotient (ISQ) | Changes in implant stability after 16 weeks (secondary stability) from baseline value measured immediately after implant placement (primary stability)
  16 weeks after implant placement, ISQ value measured by RFA device (Osstell)

CONTACTS AND LOCATIONS:
Overall Officials: Hasanain A. Al-Jumaily, C.A.B.M.S, Study Director — University of Baghdad
Locations (1):
- Mustafa Thamir Naji, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No